CLINICAL TRIAL: NCT04928729
Title: Dose Response of Pursed Lip Breathing With Diaphragmatic Breathing On Pulmonary Functions in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00879 Tayyaba Kanwal
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pursed Lip Breathing (Experimental)
  Interventions: Other: Pursed Lip Breathing
- Pursed Lip Breathing +DB (Experimental)
  Interventions: Other: Pursed Lip Breathing +DB
- Conservative care (Experimental)
  Interventions: Other: Conservative care

INTERVENTIONS:
Other: Pursed Lip Breathing — PLB with frequency of three times daily for First 3 days of week for a duration of 5-10 mins is perform.
  Arms: Pursed Lip Breathing
Other: Pursed Lip Breathing +DB — PLB+DB with frequency of three times daily for Last three days of week for a duration of 10-15 mins is perform.
  Arms: Pursed Lip Breathing +DB
Other: Conservative care — Participants will be having different dose as per tolerance 5 times daily.
  Arms: Conservative care

SUMMARY:
1. To determine the Effects of combined pursed lip breathing with diaphragmatic breathing on pulmonary functions in patient with COPD.
2. To determine the different durations of combined pursed lip breathing with diaphragmatic breathing on Pulmonary functions in patient with COPD.
3. To determine the Effects of combined pursed lip breathing with diaphragmatic breathing on quality of life in patient with COPD

DETAILED DESCRIPTION:
The technique of pursed lip breathing allow the patients to control the oxygenation and ventilation. This technique is performed by allowing the person to inspire through the nose exhale through the mouth at a slow controlled flow. This technique works by moving oxygen into your lungs and carbon dioxide out of your lungs. Pursed lip breathing (PLB) helps to slow down breathing rate and relieving shortness of breath by keeping the airways open longer. So patients can remove the air that is trapped in to the lungs.

In a recent systematic review that is published in 2018, PLB was shown to significantly improve ventilation related outcomes such as respiratory rate and minute ventilation, but not dyspnea and exercise capacity.

Diaphragmatic breathing (DB), that is also called deep breathing, this breathing is done by contracting the diaphragm, a muscle located horizontally between the thoracic cavity and abdominal cavity. During this type of breathing, air enters in to the lungs, the chest does not rise and belly expands. Diaphragmatic breathing encourages fully oxygen exchange, that is the beneficial trade of incoming oxygen for out going carbon dioxide.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed as COPD
* The intervention PLB Combine with DB
* Stable COPD Patients (Mild and Moderate on GOLD criteria) Global Initiative for Chronic Obstructive Lung Disease (GOLD)

Exclusion Criteria:

* Patients with other Pulmonary diseases.
* cardiovascular, neurological and orthopedic diseases
* Obesity, history of recent exacerbation
* Uncontrolled arterial hypertension
* Any surgical complications
* Patients with ventilatory support

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 6th week
  The COPD Assessment Test (CAT) is a questionnaire for patients with chronic obstructive pulmonary disease (COPD), which can be filled in to quantify their symptoms in the form of scores (0-40). Changes From the Baseline will be Assessed. It is categorized into four groups, that are, low(1) , medium(2), high(3) and very high(4) based on the level of effect of the disease on status of health.
Forced Expiratory Volume in 1 second (FEV1) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6th Week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 6th Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.
6 min walk test: Distance (meters) | 6th week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Modified Borg Scale of Perceived Exertion | 6th week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Pulmonology Department of DHQ Teaching Hospital, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No